CLINICAL TRIAL: NCT05385991
Title: An Open Label, Randomized, Dose and Route of Administration Comparison Phase 1 Study to Evaluate the Safety and Immunogenicity of the ACM-SARS-CoV-2-beta With ACM-CpG Vaccine Candidate (ACM-001), Administered Intramuscularly or Intranasally as a Booster Dose in Healthy Adults Aged 18 to 55 Years, Who Were Previously Vaccinated Against SARS-CoV-2.
Brief Title: Booster Dose Study to Assess the Safety and Immunogenicity of ACM-001 Administered Intramuscularly or Intranasally.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ACM Biolabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: ACM-001-01
Record Dates: First submitted 2022-05-17; First posted 2022-05-23 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-04

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — ACM-001 COVID-19 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- SARS-CoV-2 beta S vaccine arm 1 (Experimental): SARS-CoV-2 beta S vaccine Antigen dose 1, no adjuvant, IM
  Interventions: Biological: ACM-SARS-CoV-2-beta ACM-CpG vaccine candidate (ACM-001)
- SARS-CoV-2 beta S vaccine arm 2 (Experimental): SARS-CoV-2 beta S vaccine Antigen dose 1, no adjuvant, IN
  Interventions: Biological: ACM-SARS-CoV-2-beta ACM-CpG vaccine candidate (ACM-001)
- SARS-CoV-2 beta S vaccine arm 3 (Experimental): SARS-CoV-2 beta S vaccine Antigen dose 2, adjuvant dose 1, IM
  Interventions: Biological: ACM-SARS-CoV-2-beta ACM-CpG vaccine candidate (ACM-001)
- SARS-CoV-2 beta S vaccine arm 4 (Experimental): SARS-CoV-2 beta S vaccine Antigen dose 2, adjuvant dose 1, IN
  Interventions: Biological: ACM-SARS-CoV-2-beta ACM-CpG vaccine candidate (ACM-001)
- SARS-CoV-2 beta S vaccine arm 5 (Experimental): SARS-CoV-2 beta S vaccine Antigen dose 1, adjuvant dose 1, IM
  Interventions: Biological: ACM-SARS-CoV-2-beta ACM-CpG vaccine candidate (ACM-001)
- SARS-CoV-2 beta S vaccine arm 6 (Experimental): SARS-CoV-2 beta S vaccine Antigen dose 1, adjuvant dose 1, IN
  Interventions: Biological: ACM-SARS-CoV-2-beta ACM-CpG vaccine candidate (ACM-001)
- SARS-CoV-2 beta S vaccine arm 7 (Experimental): SARS-CoV-2 beta S vaccine Antigen dose 1, adjuvant dose 2, IM
  Interventions: Biological: ACM-SARS-CoV-2-beta ACM-CpG vaccine candidate (ACM-001)
- SARS-CoV-2 beta S vaccine arm 8 (Experimental): SARS-CoV-2 beta S vaccine Antigen dose 1, adjuvant dose 2, IN
  Interventions: Biological: ACM-SARS-CoV-2-beta ACM-CpG vaccine candidate (ACM-001)

INTERVENTIONS:
Biological: ACM-SARS-CoV-2-beta ACM-CpG vaccine candidate (ACM-001) — ACM-SARS-CoV-2-beta ACM-CpG vaccine candidate (ACM-001): Artificial Cell Membranes (ACM) containing recombinant SARS-CoV-2, beta- variant strain, spike protein and ACMs containing CpG adjuvant

SUMMARY:
An open label, randomized, dose comparison, sequential cohorts study design in healthy volunteers (young adults) is a frequently used design in vaccine Phase 1 studies.

ACM-001 is developed as a booster vaccine against SARS-CoV-2 after a full primary vaccination with or without 1-2 booster doses (2 or 3 or 4 doses) schedule with any registered and commercial SARS-CoV-2 vaccines.

The plan is to start with a low dosage of antigen alone, followed by a combination of antigen and adjuvant and then to progress to higher dosages to define the safety profile of the candidate vaccine as primary endpoint, and its immunogenicity as secondary endpoint.

DETAILED DESCRIPTION:
* Open label, randomized, single dose study.
* The ACM-001 vaccine will be evaluated in a single ascending dose (administered IM in 4 groups of 5 subjects and IN in 4 groups of 5 subjects), which will explore the amount of SARS-CoV-2 spike protein derived from strain B.1.351 (5 µg and 15 µg) and adjuvant CpG7909 (25 µg and 125 µg) required to provide the optimum immunogenicity and safety, as a booster dose in subjects who were previously vaccinated (two, three or four doses) against SARS-CoV-2.
* Fourty (N=40) healthy adult volunteers aged 18-55 years, will be enrolled and randomized in the IN or IM cohorts if they meet eligibility criteria at baseline. Participants who benefited from a complete 2 dose-primary vaccination with or without one or two booster dose with registered and commercial COVID-19 vaccine(s), at least 3 months prior to study vaccination (maximum 5,000 BAU/mL of anti-S Ig), with or without previous infection by COVID-19 can be enrolled in this study.
* Participants of cohorts 1,3,5 and 7 will receive an IM injection into the deltoid region, consisting of 0.4 mL per dose on Day 1. In cohorts 2, 4, 6 and 8, the vaccine will be administered IN (2 x 0.2 mL per dose) on Day 1.
* Participants will be observed closely in the research unit for at least 2 hours following vaccination.
* As from Day 30 (following completion of Day 29 visit), subjects may receive an additional (3rd or 4th or 5th) commercial SARS-CoV-2 vaccine dose.
* All subjects (having received or not a commercial dose of a SARS-CoV-2 vaccine at any point of time during their study participation) will be followed up for safety and immunogenicity on Day 85 and Day 180 visits.
* Solicited local and systemic AEs will be collected for 7 days following the vaccination using a daily reactogenicity electronic diary (eDiary). Non-serious unsolicited AEs will be collected from administration until 28 days following vaccination. Serious AEs (SAEs) and AEs of special interest (AESI; list determined by the Safety Platform for Emergency Vaccines (SPEAC; Brighton collaboration)) will be collected throughout the whole 6-month study period.
* Sentinel dosing will be applied to all cohorts for the early detection of safety signals. Two subjects will be dosed ahead of the other volunteers (at least 48 hours), with an interval of at least 2 hours between them, to ensure there are no serious acute reactions following vaccination. After global evaluation by the Investigator (or the responsible physician) and phone contact with the subjects on Day 3, and providing there are no safety concerns, the rest of the cohort (N=3) will be dosed.
* Seven-day safety data of all subjects (N=10) of a given Ag/CpG dose level will be reviewed by an independent data safety monitoring board (DSMB). The interval between the last subject receiving his/her vaccine and vaccination of three sentinel subjects with the ascending dose levels will be at least 10 days.
* On Day 1 (pre-vaccination) and on Days 8 and 29 (28 days post-vaccination), blood samples will be drawn for analysis of safety parameters.
* At all timepoints, serum and saliva samples will be collected for analysis of the humoral immune responses (IgG, IgA and neutralizing antibodies).
* The duration of the study for each subject will be approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to any study-related procedure;
2. Subjects must have received a complete primary vaccination schedule and a third and/or fourth booster dose with registered and commercial vaccine(s) against SARS-CoV-2, of which the last dose was given at least 3 months prior to study vaccination (maximum of 1,000 IU of anti-S IgG);
3. Healthy males and females, 18-55 years of age, inclusive at screening;
4. Body mass index (BMI) ≥ 18.0 and < 30.0 kg/m2;
5. Good health, based upon the results of medical history, physical examination, vital signs, laboratory profiles of both blood and urine, and according to the clinical judgement of the investigator;
6. Female participants of childbearing potential must be willing to comply with effective contraception up to 90 days after the study vaccine administration;
7. Willing to comply with the study procedures.

Exclusion Criteria:

* 1. Known immune deficiency; 2. Chronic airway disease; 3. Has experienced an acute illness, as determined by the investigator, or fever (>38.5°C) within 72 hours prior to study vaccine administration; in such case, the subject may be screened again after normalization of the temperature and/or healing of the illness; 4. Active hay fever or other active allergies involving the lower airways (bronchial and pulmonary); 5. Laboratory-confirmed PCR positive result for SARS-CoV-2 in nose/throat swab during screening; 6. Previous participation in a study to evaluate a non-registered COVID-19 vaccine within 3 months prior to study vaccination; 7. Received any other commercial vaccine within the 28 days prior to enrolment in the study, or immunization planned within 3 months after enrolment in the study (influenza vaccines are allowed up to one week before and one week after study vaccination; Exclusion criteria CONFIDENTIAL Cohort 2: 15 μg Protein (N=10), IN Cohort 4: 5 μg Protein, 25 μg CpG (N=10), IN Cohort 6: 15 μg Protein, 25 μg CpG (N=10), IN Cohort 8: 15 μg Protein, 125 μg CpG (N=10), IN ACM-001-01 Version 2.0 09 May 2022 Page 10 of 74 DocuSign Envelope ID: C34D91C3-4686-427D-BB78-CF7178216E74 CONFIDENTIAL 8. Any confirmed severe allergic reactions (urticaria, angioedema or anaphylaxis); 9. Evidence of any other active or chronic disease (hematologic, renal, hepatic, cardiovascular, neurologic, endocrinal, gastrointestinal, oncologic, pulmonary, immunologic or psychiatric disorders) or condition that could interfere with, or for which the treatment of might interfere with the conduct of the study, or that would pose an unacceptable risk to the subject in the opinion of the investigator (following a detailed medical history, physical examination, vital signs (systolic and diastolic blood pressure, and body temperature). Minor deviations from the normal range may be accepted, if judged without clinical relevance by the Investigator; 10. Clinicallysignificantabnormalities,asjudgedbytheInvestigator,in laboratory test results (including blood chemistry, hematology and urinalysis). In the case of uncertain or questionable results, tests performed during screening may be repeated before randomization to confirm eligibility or judged to be clinically irrelevant for healthy subjects; 11. Positive hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus antibody at screening; 12. Asplenia; 13. Useofanychronictreatmentwithsystemiccorticosteroids(episodic treatments with topical and intranasal corticosteroids are allowed) and immunosuppressive drugs; 14. Use of paracetamol or non-steroidal anti-inflammatory drugs (NSAIDs) within 72 hours prior to vaccination; 15. Receivedbloodproducts(transfusionsorimmunoglobulins)within3 months prior to screening, or planned administration of blood products or immunoglobulins during the study; 16. History of substance use disorder (alcohol, illegal substances), current alcohol use disorder (according to Australian guidelines: https://www.health.gov.au/news/australian-alcohol-guidelines- revised) or drug abuse; 17. Participation in an investigational drug or device study within 3 months prior to first study vaccine administration or more than 4 times a year; 18. Lossordonationofbloodover500mLwithin3months(males)or4 months (females) prior to screening or intention to donate blood or blood products during the study; 19. History of bleeding disorder (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions), significant bleeding or bruising following IM injections or venous punctures, or currently receiving anticoagulants; 20. Has body art (e.g., tattoos), skin lesions or abnormalities that could interfere with the observation of injection site reactions; ACM-001-01 Version 2.0 09 May 2022 Page 11 of 74

DocuSign Envelope ID: C34D91C3-4686-427D-BB78-CF7178216E74 Endpoints 21. Close contact with laboratory-confirmed COVID-19 cases within 10 days prior to vaccination, high risk of exposure or has an occupation with a high risk of exposure to SARS-CoV-2 (emergency response); 22. Pregnancy confirmed by a positive pregnancy test, lactation or intention to become pregnant during the study; 23. Any cancer diagnosed and/or treated within the past 5 years (except basal cell carcinoma of the skin and cervical carcinoma in situ); 24. Veins not suitable for repeated blood sampling; 25. Serious reaction, such as anaphylactic reaction, following primary COVID-19 vaccination; 26. Any known factor, condition, or disease that might interfere with treatment compliance, study conduct or interpretation of the results; 27. Sponsor employees or Investigator site personnel directly affiliated with this study, and their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted, including children of newly composed families.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-22 (Actual)

PRIMARY OUTCOMES:
Adverses events | through study completion, an average of 6 months
  Frequency, duration and intensity of solicited local AEs reported during 7 days following vaccination: injection site pain, erythema/redness (including size), and swelling/induration (including size) after IM injection, or nose pain, ear pain, runny nose, sneezing, stuffy nose and throat pain after IN administration.

SECONDARY OUTCOMES:
Immune responses | through study completion, an average of 6 months
  Humoral and mucosal immune responses

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (6):
  - Paratus Research Central Coast, Kanwal, New South Wales
  - Paratus Research Sydney, Sydney, New South Wales
  - Paratus research Brisbane, Brisbane, Queensland
  - Paratus research Canberra, Canberra
  - Emeritus Research Melbourne, Melbourne
  - Emeritus Research Sydney, Sydney

REFERENCES:
- [Derived] Dress RJ, Ho WW, Ho V, Lam JH, Decaillot FM, Sinsinbar G, Soo J, Rengasamy G, Khan AK, Cornell TA, Chia TW, Venkataraman S, Nallani M, Ginhoux F. A Novel Polymersome Nanocarrier Promotes Anti-Tumour Immunity by Improved Priming of CD8 + T Cells. Immunology. 2025 May;175(1):21-35. doi: 10.1111/imm.13903. Epub 2025 Jan 28. PMID 39873184
- [Derived] Nakahashi-Ouchida R, Fujihashi K, Kurashima Y, Yuki Y, Kiyono H. Nasal vaccines: solutions for respiratory infectious diseases. Trends Mol Med. 2023 Feb;29(2):124-140. doi: 10.1016/j.molmed.2022.10.009. Epub 2022 Nov 23. PMID 36435633
- [Derived] Lam JH, Shivhare D, Chia TW, Chew SL, Sinsinbar G, Aw TY, Wong S, Venkataraman S, Lim FWI, Vandepapeliere P, Nallani M. Artificial Cell Membrane Polymersome-Based Intranasal Beta Spike Formulation as a Second Generation Covid-19 Vaccine. ACS Nano. 2022 Oct 25;16(10):16757-16775. doi: 10.1021/acsnano.2c06350. Epub 2022 Oct 12. PMID 36223228